CLINICAL TRIAL: NCT04716933
Title: A Phase 3 Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of Pemetrexed + Platinum Chemotherapy + Pembrolizumab (MK-3475) With or Without Lenvatinib (E7080/MK-7902) as First-line Intervention in Participants With Metastatic Nonsquamous Non-small Cell Lung Cancer (LEAP-006)
Brief Title: Safety and Efficacy Study of Pemetrexed + Platinum Chemotherapy + Pembrolizumab (MK-3475) With or Without Lenvatinib (MK-7902/E7080) as First-line Intervention in Adults With Metastatic Nonsquamous Non-small Cell Lung Cancer (MK-7902-006/E7080-G000-315/LEAP-006)-China Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7902-006 China Extension; MK-7902-006 (Other: Merck); E7080-G000-315 (Other: Eisai Protocol Number); LEAP-006 (Other: MSD)
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Nonsquamous Non-small Cell Lung Cancer
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death-ligand 1 (PD-L1, PDL1); programmed cell death-ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Cisplatin; Pemetrexed; lenvatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib (Experimental): Participants receive carboplatin Area Under Curve 5 mg/mL/min (AUC5) or cisplatin 75 mg/m^2 via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) for 4 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pembrolizumab via IV infusion Q3W for up to 35 cycles (up to 2 years) PLUS lenvatinib via oral capsule once daily.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Lenvatinib
- Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo (Placebo Comparator): Participants receive carboplatin AUC5 or cisplatin 75 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pembrolizumab via IV infusion Q3W for up to 35 cycles (up to 2 years) PLUS (Part 2 only) placebo matching lenvatinib via oral capsule once daily.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Placebo matching lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion Q3W
  Other Names: MK-3475
Drug: Carboplatin — IV infusion Q3W
Drug: Cisplatin — IV infusion Q3W
Drug: Pemetrexed — IV infusion Q3W
Drug: Lenvatinib — Oral capsule once daily
  Other Names: MK-7902; E7080
  Arms: Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib
Drug: Placebo matching lenvatinib — Oral capsule once daily
  Arms: Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of pemetrexed+platinum chemotherapy+pembrolizumab (MK-3475) with or without lenvatinib (MK-7902/E7080) as first-line intervention in adults from mainland China with metastatic nonsquamous non-small cell lung cancer.

The primary study hypotheses state that: 1) the combination of lenvatinib+platinum doublet chemotherapy+pembrolizumab prolongs Progression-free Survival (PFS) as assessed by blinded independent central review (BICR) per modified Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST 1.1) compared to matching placebo+platinum doublet chemotherapy+pembrolizumab, and 2) the combination of lenvatinib+platinum doublet chemotherapy+pembrolizumab prolongs Overall Survival (OS) compared to matching placebo+platinum doublet chemotherapy + pembrolizumab.

DETAILED DESCRIPTION:
The China extension study will include participants previously enrolled in mainland China for the global study for MK-7902-006 (NCT03829319) plus those enrolled in mainland China as part of the China extension enrollment period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of Stage IV (American Joint Committee on Cancer [AJCC], version 8 or current version) nonsquamous NSCLC.
* Confirmation that Epidermal Growth Factor Receptor (EGFR), ALK Receptor Tyrosine Kinase (ALK), or ROS1 Receptor Tyrosine Kinase (ROS1)-directed therapy is not indicated as primary treatment (documentation of absence of tumor-activating EGFR mutations AND absence of ALK and ROS1 gene rearrangements OR presence of a Kirsten Rat Sarcoma (KRAS) gene mutation).
* Have measurable disease based on RECIST 1.1. Note: Lesions that appear measurable, but are situated in a previously irradiated area, can be considered measurable (eligible for selection as target lesions) if they have shown documented growth since the completion of radiation.
* Provided an evaluable archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion (that was not previously irradiated) for central PD-L1 testing.
* Life expectancy of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to the first dose of study intervention but before randomization.
* Male participants must agree to use contraception during the treatment period and for at least 120 days after the last dose of pembrolizumab and/or lenvatinib/matching placebo and up to 180 days after the last dose of chemotherapeutic agents. A male participant must also agree to the following: 1) abstinence from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR 2) agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant, unless confirmed to be azoospermic (vasectomized or secondary to medical cause). Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.
* Female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: 1) not a WOCBP OR 2) a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 120 days after the last dose of study intervention.
* Adequate organ function.
* Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg and no change in antihypertensive medications within 1 week prior to randomization. Note: Participants must not have a history of uncontrolled or poorly-controlled hypertension, defined as >150/90 mm Hg for >4 weeks despite standard medical management.

Exclusion Criteria:

* Known untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, clinically stable, and have not required steroids for at least 14 days prior to the first dose of study intervention.
* History of (noninfectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease.
* Radiographic evidence of major blood vessel invasion/infiltration.
* Known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for at least 3 years since initiation of that therapy. Note: The time requirement also does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention.
* Has had allogeneic tissue/solid organ transplant.
* Known history of human immunodeficiency virus (HIV) infection. HIV testing is not required unless mandated by the local health authority.
* Known history of Hepatitis B or active Hepatitis C. No testing for Hepatitis B or Hepatitis C is required unless mandated by the local health authority.
* History of a gastrointestinal condition or procedure that in the opinion of the investigator may affect oral drug absorption.
* Active hemoptysis (at least 0.5 teaspoon of bright red blood) within 2 weeks prior to the first dose of study intervention.
* Significant cardiovascular impairment within 12 months prior to the first dose of study intervention, including history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, cerebrovascular accident (CVA)/stroke, or cardiac arrhythmia associated with hemodynamic instability.
* Known history of active tuberculosis.
* Active infection requiring systemic therapy.
* Has not recovered adequately from any toxicity and/or complication from major surgery prior to the first dose of study intervention.
* Previously had a severe hypersensitivity reaction to treatment with a monoclonal antibody or has a known sensitivity to any component of lenvatinib or pembrolizumab, or as applicable, carboplatin, cisplatin, or pemetrexed.
* Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of pembrolizumab and/or lenvatinib/matching placebo and up to 180 days after last dose of chemotherapeutic agents.
* Received prior systemic chemotherapy or other targeted or biological antineoplastic therapy for their metastatic NSCLC. Note: Prior treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic NSCLC.
* Received prior treatment with pembrolizumab or any other anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2 agent, with lenvatinib or any other receptor tyrosine kinase inhibitor (RTKi), or with an agent directed to another stimulatory or co-inhibitory T cell receptor.
* Received radiotherapy within 14 days prior to the first dose of study intervention or received lung radiation therapy of >30 Gy within 6 months prior to the first dose of study intervention. Note: Participants must have recovered from all radiation-related toxicities to Grade ≤1, not required corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Received systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) within 7 days prior to the first dose of study intervention.
* Received a live vaccine within 30 days prior to the first dose of study intervention.
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has a prolongation of QTc interval (calculated using Fridericia's formula) of >480 msec
* Left ventricular ejection fraction (LVEF) below the institutional (or local laboratory) normal range as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO).
* Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (19):
- China (19):
  - Peking Union Medical College Hospital ( Site 0108), Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Science ( Site 0117), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0120), Beijing, Beijing Municipality
  - The Second Hospital Affiliated to AMU ( Site 0119), Chongqing, Chongqing Municipality
  - First Affiliated Hospital of The Third Military Medical University ( Site 0118), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0102), Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital ( Site 0121), Guangzhou, Guangdong
  - The Third Affiliated Hospital of Harbin Medical University ( Site 0100), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 0112), Zhengzhou, Henan
  - Wuhan Union Hospital ( Site 0123), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 0122), Wuhan, Hubei
  - Zhongshan Hospital Fudan University ( Site 0103), Shanghai, Hunan
  - Jilin Cancer Hospital ( Site 0115), Changchun, Jilin
  - Shanghai Pulmonary Hospital ( Site 0101), Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0111), Tianjin, Tianjin Municipality
  - Cancer Hospital Affiliated to Xinjiang Medical University ( Site 0110), Urumuqi, Xinjiang
  - The First Affiliated Hospital Zhejiang University ( Site 0109), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0113), Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 0124), Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 201 Chinese participants were randomized and received treatment as a part of global study [NCT03829319; n=761] or to the extension portion.
  No participants from China were randomized to Part 1.
Groups:
- Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib: Participants received carboplatin Area Under Curve 5 mg/mL/min (AUC5) or cisplatin 75 mg/m^2 via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) for 4 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pembrolizumab via IV infusion Q3W for up to 35 cycles (up to 2 years) PLUS lenvatinib via oral capsule once daily.
- Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo: Participants received carboplatin AUC5 or cisplatin 75 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pembrolizumab via IV infusion Q3W for up to 35 cycles (up to 2 years) PLUS (Part 2 only) placebo matching lenvatinib via oral capsule once daily.
Period: Overall Study
Arm/Group | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo
Started | 101 | 100
Completed | 0 | 0
Not Completed | 101 | 100
Not completed — Sponsor Decision | 36 | 33
Not completed — Death | 65 | 67

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo | Total
Number analyzed (Participants) | 101 | 100 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (8.6) | 60.9 (8.2) | 59.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 78 | 74 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 101 | 100 | 201
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 101 | 100 | 201
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG = 0 | 20 | 21 | 41
    ECOG = 1 | 81 | 79 | 160
Programmed Cell Death Ligand 1 (PD-L1) Status at Baseline [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Randomization of participants in the study was stratified by PD-L1 tumor proportion score (TPS) at baseline (< 50% or ≥ 50%). Higher percentages of PD-L1 TPS staining correspond to higher positivity of PD-L1 on a tumor.
  Participants
    TPS = < 50% | 77 | 81 | 158
    TPS = ≥ 50% | 24 | 18 | 42
    Not Evaluable | 0 | 1 | 1
Geographic Region [Count of Participants; unit: Participants] — Randomization of participants in this study was stratified by geographic region of the enrolling site (East Asia or non-East Asia).
  Participants
    East Asia | 101 | 100 | 201
    Non-East Asia | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS is defined as the time from date of randomization to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurred first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. Data are from the product-limit (Kaplan-Meier) method for censored data. PFS as assessed by blinded independent central review (BICR) per RECIST 1.1 is presented.
Time Frame: Up to approximately 43 months
Population: All Chinese participants who were randomized to the global study (NCT03829319) or to the extension portion that were evaluable for response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo
Number analyzed (Participants) | 101 | 100
Months | 15.3 [12.2 to 19.6] | 9.2 [8.2 to 12.5]
Statistical Analysis 1: Comparison: Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib vs Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo; Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Test type: Other; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.48 to 0.97]

2. Primary Outcome: Part 2: Overall Survival (OS)
Description: OS is defined as the time from randomization to the time of death from any cause. OS is presented.
Time Frame: Up to approximately 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo
Number analyzed (Participants) | 101 | 100
Months | 26.6 [22.2 to 35.0] | 22.0 [16.6 to 24.8]
Statistical Analysis 1: Comparison: Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib vs Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo; Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Test type: Other; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.54 to 1.12]

3. Secondary Outcome: Part 2: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. ORR as assessed per modified RECIST 1.1 will be presented.
Time Frame: Up to approximately 57 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo
Number analyzed (Participants) | 101 | 100
Percentage of participants | 70.3 [60.4 to 79.0] | 59.0 [48.7 to 68.7]
Statistical Analysis 1: Comparison: Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib vs Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo; Comparision based on unstratified Miettinen & Nurminen method; Test type: Other; Percent Difference = 11.3, 95% CI 2-sided [-2.0 to 24.2]

4. Secondary Outcome: Part 2: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: For participants who demonstrated CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), DOR is defined as the time from the first documented evidence of CR or PR until PD or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, or death from any cause, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. DOR as assessed per modified RECIST 1.1 will be presented.
Time Frame: Up to approximately 57 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo
Number analyzed (Participants) | 62 | 51
Months | 17.0 [12.6 to 23.6] | 12.5 [6.7 to 27.5]

5. Secondary Outcome: Part 2: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced one of more adverse events during Part 2 of this study were presented.
Time Frame: Up to approximately 42 months
Population: All Chinese participants who were randomized to the global study (NCT03829319) or to the extension portion who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo
Number analyzed (Participants) | 101 | 100
Participants | 101 | 100

6. Secondary Outcome: Part 2: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment during Part 2 of this study were presented.
Time Frame: Up to approximately 42 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo
Number analyzed (Participants) | 101 | 100
Participants | 42 | 21

ADVERSE EVENTS:
Time Frame: Up to approximately 42 months for first course and up to approximately 57 months for second course. All-cause mortality (ACM): Up to approximately 57 months for first and second course.
Description: All-cause mortality includes all randomized participants. Safety includes participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE, unless related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment were excluded as AEs
Groups:
- Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo(Second Course): Qualified participants who completed the first course of pembrolizumab plus chemotherapy plus lenvatinib for up to 35 cycles (up to 2 years), but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q2W for up to ~1 year. Participants previously receiving placebo could continue receiving placebo at investigator's discretion.
Arm/Group | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo(Second Course)
All-Cause Mortality (participants affected / at risk) | 65/101 | 67/100 | 0/2
Serious Adverse Events (participants affected / at risk) | 67/101 | 53/100 | 1/2
Other Adverse Events (participants affected / at risk) | 100/101 | 99/100 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib (N=101) | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo (N=100) | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo(Second Course) (N=2)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 3 (4) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal haematoma (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric mucosal lesion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 3 (3) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 12 (13) | 16 (18) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 6 (6) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 4 (5) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 4 (4) | 0 (0)
Platelet count decreased (Investigations) | 7 (8) | 4 (4) | 0 (0)
White blood cell count decreased (Investigations) | 3 (4) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal tubular injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis herpetiformis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib (N=101) | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo (N=100) | Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo(Second Course) (N=2)
Anaemia (Blood and lymphatic system disorders) | 84 (266) | 82 (224) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 5 (9) | 10 (14) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 6 (8) | 7 (7) | 0 (0)
Hypothyroidism (Endocrine disorders) | 25 (43) | 14 (17) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 6 (9) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 9 (11) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 26 (44) | 41 (55) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 19 (36) | 13 (16) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 9 (14) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 14 (14) | 7 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 34 (91) | 35 (67) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (9) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 10 (14) | 6 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 23 (32) | 19 (24) | 0 (0)
Asthenia (General disorders) | 15 (21) | 10 (19) | 0 (0)
Chest discomfort (General disorders) | 10 (11) | 9 (9) | 0 (0)
Chest pain (General disorders) | 5 (6) | 13 (15) | 0 (0)
Fatigue (General disorders) | 23 (27) | 17 (27) | 0 (0)
Malaise (General disorders) | 5 (7) | 6 (6) | 0 (0)
Oedema peripheral (General disorders) | 8 (11) | 12 (26) | 0 (0)
Pyrexia (General disorders) | 17 (31) | 17 (21) | 1 (1)
COVID-19 (Infections and infestations) | 12 (14) | 10 (10) | 0 (0)
Pneumonia (Infections and infestations) | 11 (13) | 6 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (24) | 13 (18) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (6) | 7 (11) | 0 (0)
Alanine aminotransferase increased (Investigations) | 63 (191) | 58 (183) | 0 (0)
Amylase increased (Investigations) | 21 (35) | 18 (31) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 67 (226) | 61 (188) | 0 (0)
Bilirubin conjugated increased (Investigations) | 9 (13) | 5 (7) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 22 (44) | 18 (29) | 0 (0)
Blood bilirubin increased (Investigations) | 14 (20) | 7 (10) | 0 (0)
Blood creatinine increased (Investigations) | 28 (65) | 22 (45) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 16 (46) | 10 (16) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 14 (20) | 3 (5) | 0 (0)
Blood urea increased (Investigations) | 6 (8) | 4 (5) | 0 (0)
Blood uric acid increased (Investigations) | 7 (14) | 5 (7) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 7 (9) | 6 (8) | 0 (0)
Fibrin D dimer increased (Investigations) | 11 (11) | 3 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 37 (69) | 34 (51) | 0 (0)
Lipase increased (Investigations) | 14 (21) | 11 (12) | 0 (0)
Lymphocyte count decreased (Investigations) | 21 (52) | 12 (28) | 0 (0)
Neutrophil count decreased (Investigations) | 83 (401) | 74 (326) | 0 (0)
Platelet count decreased (Investigations) | 65 (248) | 47 (140) | 0 (0)
Urinary occult blood positive (Investigations) | 7 (9) | 6 (8) | 1 (1)
Weight decreased (Investigations) | 29 (37) | 14 (16) | 0 (0)
Weight increased (Investigations) | 20 (30) | 7 (8) | 0 (0)
White blood cell count decreased (Investigations) | 78 (366) | 70 (293) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 38 (89) | 44 (78) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 26 (61) | 16 (43) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (18) | 4 (7) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 8 (10) | 2 (7) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12 (73) | 13 (46) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 15 (31) | 13 (35) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 34 (78) | 25 (62) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 14 (27) | 7 (19) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 9 (22) | 7 (8) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (40) | 18 (25) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 25 (51) | 15 (26) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 12 (27) | 5 (11) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 12 (14) | 9 (20) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 14 (18) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (17) | 9 (10) | 0 (0)
Dizziness (Nervous system disorders) | 10 (11) | 13 (21) | 0 (0)
Headache (Nervous system disorders) | 8 (10) | 9 (13) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (10) | 13 (22) | 0 (0)
Albuminuria (Renal and urinary disorders) | 8 (27) | 4 (6) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (19) | 7 (12) | 0 (0)
Proteinuria (Renal and urinary disorders) | 33 (75) | 23 (35) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (24) | 14 (18) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 10 (10) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (28) | 3 (4) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (5) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 6 (11) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 11 (11) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 10 (18) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 19 (28) | 14 (15) | 0 (0)
Hypertension (Vascular disorders) | 34 (51) | 5 (6) | 1 (1)
Degenerative aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT04716933/Prot_SAP_002.pdf